CLINICAL TRIAL: NCT06204497
Title: The Safety and Efficiency of Stent-based Diverting Technique Versus Ileostomy in Rectal Cancer Patients: A Prospective, Multicenter, Open-label, Non-inferiority, Randomized Controlled Study
Brief Title: The Safety and Efficiency of Stent-based Diverting Technique Versus Ileostomy in Rectal Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xiujun Cai, Director, Head of General Surgery, Principal Investigator, Clinical Professor, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRRSH.SDT
Record Dates: First submitted 2023-12-12; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Rectal Neoplasms
Keywords: Stent-based diverting technique; Ileostomy; Complication; Anastomotic leakage
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: The patients who were enrolled will either undergo ileostomy or SDT after the removal of the rectal tumor, which will be decided by chance.
Who Masked: Outcomes Assessor
Masking Description: The masking in this study is inappropriate because the patients in the SDT group do not have an abdominal stoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent-based Diverting Technique (Experimental): For Stent-based Diverting Technique, the small intestine measuring 15 cm from the ileocecal junction was pulled out through the median incision in the lower abdomen. After a length-wise incision was established in the mesenteric margin of the small intestine, the degradable stent was implanted, and the intestine was sutured. Then, the stent was held in place using an external tie around the bowel. Next, a mushroom-like tube (28 Fr) was placed into the intestine proximal (5-10 cm) to the aforementioned stent. The other side of the mushroom-like tube was inserted through the right lower abdominal wall and connected with a drainage bag. An abdominal drainage tube, or an anal tube, if necessary, was inserted in the proper location prior to the closure of the incision and the abdominal cavity. Abdominal X-ray was routinely performed every week to detect stent degradation, and the mushroom-like tube (28 Fr) was removed two days after stent degradation.
  Interventions: Procedure: Stent-based Diverting Technique
- Ileostomy (Active Comparator): There will be an ileostomy for the control group. An incision with a diameter of 2 cm will be performed in the lower abdomen, and layers will be separated into the abdominal cavity. The intestine, 20cm to the ileocecal juction under laparoscopic vision, will be pulled out. The anterior sheath of the rectus abdominis and the serous layer of the intestine will be sutured with an absorbable line. Then, the middle point of the mesangial margin of the intestine will be transected, and the intestine will be fixed on the skin. No volvulus or angular formation of the intestine should be confirmed laparoscopically.
  Interventions: Procedure: Stent-based Diverting Technique

INTERVENTIONS:
Procedure: Stent-based Diverting Technique — The stent-based diverting technique (SDT) contains two parts to achieve feces diversion One is a degradable solid intestinal stent to be implanted 20 cm from the terminal ileum and could be gradually degraded within 3-4 weeks. Another part is a drainage tube to be placed at the proximal 5-10 cm of the aforementioned stent. Given this SDT, intestinal contents could be diverted through the drainage tube, and the stent prevents the feces from entering the distal intestinal. After removing the drainage tube after 3-4 weeks, intestinal contents will freely access the distal intestinal space following the degradation of the stent. For patients, stoma reversal is avoided.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficiency of stent-based tiverting technique (SDT) versus ileostomy in rectal cancer patients. After the removal of the rectal tumor, participants who are at high risk for anastomotic leakage will either undergo SDT or ileostomies. Researchers will compare SDT to see if SDT could help patients save hospital stays, lower medical costs, and enhance their quality of life, and not alternatively avoid defunction stoma.

DETAILED DESCRIPTION:
In patients with rectal cancer who have a high risk of anastomotic leakage, we aim to compare the safety and effectiveness of SDT versus ileostomy in this study. The primary endpoint of the study was severe complications that occurred within 90 days of the surgery. The secondary endpoints included total complications, the incidence of coloanal anastomotic leakage (Grade B/C), postoperative hospital stay and cost, and postoperative quality of life evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal adenocarcinoma confirmed pathologically.
2. Rectal cancer patients with high-risk of anastomotic leakage(AL).
3. Age from over 18 to under 80 years.
4. Performance status of 0/1 on ECOG (Eastern Cooperative Oncology Group) scale.
5. ASA (American Society of Anesthesiology) score class I, II, or III.
6. Written informed consent.

Definition of high-risk of AL (one of them):

1. Preoperative body mass index (BMI) ≥30 kg/m2;
2. Long-term use of glucocorticoids before surgery (≥2 weeks);
3. Poor general condition: Preoperative serum albumin was less than 30.0g/L after supportive treatment; or Preoperative renal replacement therapy (blood purification/hemodialysis) is required; or diabetes;
4. Preoperative neoadjuvant radiotherapy;
5. Distance between tumor and anal anus (baseline MRI) ≤7cm
6. The number of stapler used to cut the rectum during the operation ≥3; or the defect of anastomosis is observed; or Intraoperative leak test was positive.

Exclusion Criteria:

1. History of previous rectectomy, except endoscopic mucosal resection or endoscopic submucosal dissection.
2. Familial Adenomatosis Polyposis Coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active colitis ulcerosa.
3. History of unstable angina, myocardial infarction, cerebrovascular accident within the past six months.
4. Groups who are particularly vulnerable include those who suffer from mental disease, cognitive impairment, severe illness, adolescents, illiterates, women during pregnancy or breast-feeding, etc.
5. Patients with severe complications who do not tolerate surgery or need emergency surgery due to complication (bleeding, obstruction or perforation)
6. Unable ot radical resection, or underwent Miles or Hartmann or TaTME procedure, or requirement of simultaneous surgery for other disease (except the gallblader or appendix due to benign lesion).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe complications within 90-day | Study group, from SDT to postoperative 90 days, Control group, from ileostomy to postoperative 90 days of reversal of stoma.
  Clavein-Dindo≥III

SECONDARY OUTCOMES:
Total complications | Study group, from SDT to postoperative 90 days; Control group, from ileostomy, plus interval time before stoma reversal, to postoperative 90 days of reversal of stoma
  Clavein-Dindo I to V
Clinical anastomotic leakage | Study group, from SDT to postoperative 90 days; Control group, from ileostomy, plus interval time before stoma reversal, to postoperative 90 days of reversal of stoma
  Grade B or Grade C
Postoperative hospital stay | Study group, from SDT to discharge, and adding second postoperative hospital stay if the patient received the ileostomy. Control group, from ileostomy to discharge and from stoma reversal to discharge，up to six months for both group
  Postoperative hospital stay after SDT or ileostomy or reversal of stoma
Total medical Costs | From first admission to end of follow-up or date of death from any cause, whichever came first, assessed up to six months for both group
  Including medical costs, surgery costs and other costs
Quality of life evaluation | Study group, 90 days after SDT; Control group, 90 days after ileostomy
  SF-8 scale

CONTACTS AND LOCATIONS:
Overall Officials: XiuJun Cai, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (20):
- China (20):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Peking University, Beijing, Beijing Municipality
  - Peking Union Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospita, Beijing, Beijing Municipality
  - Fujian Union Hospital, Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South Universit, Changsha, Hunan
  - The First Affiliated Hospital, Jilin University, Jilin, Jilin
  - Shengjing Hospital, China Medical University, Shenyang, Liaoning
  - The Affiliated Hospital, Qingdao University, Qingdao, Shandong
  - Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality
  - ChangHai Hospital, The Second Military Medical University, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, University of Electronic Science and Technology of China, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Ningbo University, Ningbo, Zhejiang
  - The Second Affiliated Hospital, Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
The data are available from the Principal Investigator upon reasonable request.

REFERENCES:
- [Background] Bonjer HJ, Deijen CL, Abis GA, Cuesta MA, van der Pas MH, de Lange-de Klerk ES, Lacy AM, Bemelman WA, Andersson J, Angenete E, Rosenberg J, Fuerst A, Haglind E; COLOR II Study Group. A randomized trial of laparoscopic versus open surgery for rectal cancer. N Engl J Med. 2015 Apr 2;372(14):1324-32. doi: 10.1056/NEJMoa1414882. PMID 25830422
- [Background] Sparreboom CL, van Groningen JT, Lingsma HF, Wouters MWJM, Menon AG, Kleinrensink GJ, Jeekel J, Lange JF; Dutch ColoRectal Audit group. Different Risk Factors for Early and Late Colorectal Anastomotic Leakage in a Nationwide Audit. Dis Colon Rectum. 2018 Nov;61(11):1258-1266. doi: 10.1097/DCR.0000000000001202. PMID 30239395
- [Background] Borstlap WAA, Westerduin E, Aukema TS, Bemelman WA, Tanis PJ; Dutch Snapshot Research Group. Anastomotic Leakage and Chronic Presacral Sinus Formation After Low Anterior Resection: Results From a Large Cross-sectional Study. Ann Surg. 2017 Nov;266(5):870-877. doi: 10.1097/SLA.0000000000002429. PMID 28746154
- [Background] Zhou S, Zhou H, Zheng Z, Liang J, Zhou Z, Wang X. Predictive risk factors for anastomotic leakage after anterior resection of rectal cancer in elderly patients over 80 years old: an analysis of 288 consecutive patients. World J Surg Oncol. 2019 Jun 29;17(1):112. doi: 10.1186/s12957-019-1655-z. PMID 31255181
- [Background] Wu J, Lu AD, Zhang LP, Zuo YX, Jia YP. [Study of clinical outcome and prognosis in pediatric core binding factor-acute myeloid leukemia]. Zhonghua Xue Ye Xue Za Zhi. 2019 Jan 14;40(1):52-57. doi: 10.3760/cma.j.issn.0253-2727.2019.01.010. Chinese. PMID 30704229
- [Background] Chen H, Cai HK, Tang YH. An updated meta-analysis of transanal drainage tube for prevention of anastomotic leak in anterior resection for rectal cancer. Surg Oncol. 2018 Sep;27(3):333-340. doi: 10.1016/j.suronc.2018.05.018. Epub 2018 May 22. PMID 30217286
- [Background] Mrak K, Uranitsch S, Pedross F, Heuberger A, Klingler A, Jagoditsch M, Weihs D, Eberl T, Tschmelitsch J. Diverting ileostomy versus no diversion after low anterior resection for rectal cancer: A prospective, randomized, multicenter trial. Surgery. 2016 Apr;159(4):1129-39. doi: 10.1016/j.surg.2015.11.006. Epub 2015 Dec 17. PMID 26706610
- [Background] Rao S, Guren MG, Khan K, Brown G, Renehan AG, Steigen SE, Deutsch E, Martinelli E, Arnold D; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Anal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up☆. Ann Oncol. 2021 Sep;32(9):1087-1100. doi: 10.1016/j.annonc.2021.06.015. Epub 2021 Jun 24. No abstract available. PMID 34175386
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914